CLINICAL TRIAL: NCT04471077
Title: Association Between Outcomes of Bariatric Surgery and Preoperative Gastrointestinal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Stefura, Reasearch Associate, PhD student at 2nd Department of General Surgery, Principal Investigator, Medical Doctor, Jagiellonian University
Other Study IDs: 1072.6120.196.2018
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Favorable outcome of bariatric surgery: Excess weight loss above 50%
  Interventions: Procedure: bariatric surgery
- Unfavorable outcome of bariatric surgery: Excess weight loss below 50%
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — (Laparoscopic Sleeve Gastrectomy, laparoscopic Roux-en-Y gastric bypass)

SUMMARY:
Purpose The aim of this study was to analyze the microbiota of patients undergoing LSG or LRYGB on three levels of gastrointestinal tract, using oral swab and stool sample. We compared samples from patients achieving favorable outcomes in terms of weight-loss with patients, who did not respond optimally to the bariatric operation.

Materials and methods Design This prospective cohort study was conducted in one academic, teaching hospital. The recommendations of the Metabolic and Bariatric Surgery Section of the Polish Surgical Society were used as indication for surgery, that is: Body Mass Index (BMI) ≥35 kg/m2 with obesity-related comorbidities or BMI ≥40 kg/m2 .

Analysis and endpoints Primary endpoint was to determine the difference in microbiota present in oral cavity and large intestine between patients ing Group 1 and Group 2. Secondary endpoint was to compare the results of microbiota analysis between LSG and LRYGB.

ELIGIBILITY:
Inclusion Criteria:

* informed consent to participate in the study, meeting the eligibility criteria for bariatric treatment, either for LSG or LRYGB.

Exclusion Criteria:

* type 1 or type 2 diabetes, treatment with antibiotics within 30 days prior to gathering microbiological material, treatment with probiotics within 30 days prior to gathering microbiological material, gastrointestinal infections, inflammatory bowel disease, thyroid diseases, cancer (especially the digestive tract), immunodeficiency.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators included patients undergoing surgical treatment for morbid obesity.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of microbiota in oral cavity | 6 months
Change of microbiota in large intestine | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No
We are not planing to share data.